CLINICAL TRIAL: NCT04575766
Title: A Phase 1 Study of FT-7051 in Men With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of FT-7051 in Men With MCRPC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 7051-ONC-101
Record Dates: First submitted 2020-09-24; First posted 2020-10-05 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Metastatic Castration-resistant Prostate Cancer; Prostate cancer; Urogenital disease; Prostatic disease; Hormone antagonists; Hormones, hormone substitutes; FT-7051
MeSH Terms: conditions — Prostatic Neoplasms; Urogenital Diseases; Prostatic Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation study of FT-7051 (Experimental)
  Interventions: Drug: FT-7051

INTERVENTIONS:
Drug: FT-7051 — Dose levels: Dose Level -1 through Dose Level 7, assigned per the protocol using a BOIN design. Additional dose levels may be explored as applicable.
  Capsules available in strengths of 10mg, 25mg, and 100 mg that are orally administered per the protocol frequency and dose level.

SUMMARY:
This is a Phase 1, open-label study that will evaluate the safety and tolerability of FT-7051 and determine the recommended Phase 2 dose (RP2D) as well as pharmacokinetics (PK), preliminary anti-tumor activity, and pharmacodynamics (PD) of FT-7051 in men with metastatic castration-resistant prostate cancer who have progressed despite prior therapy and had been treated with at least one potent anti-androgen therapy.

The starting dose, 25 mg once daily (QD), of FT-7051 administered discontinuously (21 days on/7 days off) in 28-day cycles.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosis of progressive metastatic castration-resistant prostate cancer (mCRPC)
* Previously failed at least one potent anti-androgen therapy
* Castrate levels of serum testosterone
* ECOG performance status 0-2
* Adequate bone marrow function
* Adequate kidney, heart and liver function

Exclusion Criteria:

* Prior solid organ transplant
* Prior treatment with small molecules including chemotherapy, antibody, or other experimental anticancer therapeutic within 4 weeks of first dose of study treatment
* Prior radiation therapy within 4 weeks prior to initiation of study treatment (including radiofrequency ablation)
* Prior androgen antagonist therapy (enzalutamide, apalutamide, abiraterone acetate, or darolutamide) within 2 weeks
* Prior radium-223 therapy within 6 weeks
* Symptomatic, untreated or actively progressing central nervous system (CNS) metastasis
* Unstable or severe, uncontrolled medical condition (e.g., unstable cardiac function, unstable pulmonary condition including pneumonitis and/or interstitial lung disease, uncontrolled diabetes, active or uncontrolled infection requiring systemic therapy) or any important medical illness or abnormal laboratory finding that would, in the Investigator's judgement, increase the risk to the patient associated with participation in the study
* Concomitant medications that cause Torsades de Pointes that have not reached steady state before first dose of the study drug
* Concomitant medications that are strong inhibitors or inducers of CYP3A4 or an inhibitor of P-gp
* History of infection with human immunodeficiency virus (HIV)
* Active infection with hepatitis B, or hepatitis C virus

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Within first 4 weeks of treatment
Serious adverse events (SAEs) and clinically relevant adverse events (AEs) | The treatment duration, predicted average 26 weeks
Incidence of clinical laboratory abnormalities as assessed by CTCAE v5.0 | The treatment duration, predicted average 26 weeks

SECONDARY OUTCOMES:
Prostate-specific antigen (PSA): Percent Change from Baseline | 12 weeks
Prostate-specific antigen (PSA): Maximum Decrease from Baseline | The treatment duration, predicted average 26 weeks
Prostate-specific antigen (PSA): Time to Progression | The treatment duration, predicted average 26 weeks
Time to radiographic progression (rTTP) | The treatment duration, predicted average 26 weeks
Overall response rate: radiographic response rate | The treatment duration, predicted average 26 weeks
Complete response rate | The treatment duration, predicted average 26 weeks
Area under the plasma concentration versus time curve (AUC) | Blood samples for PK analysis collected at multiple visits during the first 90 days of treatment
Peak Plasma Concentration (Cmax) | Blood samples for PK analysis collected at multiple visits during the first 90 days of treatment
Time of peak plasma concentration (Tmax) | Blood samples for PK analysis collected at multiple visits during the first 90 days of treatment
Terminal elimination half-life (T 1/2) | Blood samples for PK analysis collected at multiple visits during the first 90 days of treatment
Apparent plasma clearance (CL/F) | Blood samples for PK analysis collected at multiple visits during the first 90 days of treatment
Apparent volume of distribution (Vd/F) | Blood samples for PK analysis collected at multiple visits during the first 90 days of treatment
Model-based estimate of change from baseline QT interval corrected using Fridericia's correction formula (QTcF) and 90% confidence interval at the estimated Cmax | Electrocardiogram collected at multiple timepoints during the first 45 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Emma Barrett, MD, Study Director — Novo Nordisk A/S
Locations (8):
- United States (8):
  - HonorHealth, Scottsdale, Arizona
  - University of Colorado Health, Aurora, Colorado
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Duke University Health System, Durham, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina

REFERENCES:
- [Derived] Caligiuri M, Williams GL, Castro J, Battalagine L, Wilker E, Yao L, Schiller S, Toms A, Li P, Pardo E, Graves B, Azofeifa J, Chicas A, Herbertz T, Lai M, Basken J, Wood KW, Xu Q, Guichard SM. FT-6876, a Potent and Selective Inhibitor of CBP/p300, is Active in Preclinical Models of Androgen Receptor-Positive Breast Cancer. Target Oncol. 2023 Mar;18(2):269-285. doi: 10.1007/s11523-023-00949-7. Epub 2023 Feb 24. PMID 36826464